CLINICAL TRIAL: NCT03839056
Title: Comparative Study of the Combination of Different Modes of Administration of Local Anesthetics in Labor Analgesia
Status: Completed | Type: Observational
Sponsor: Marian Daras (Other)
Collaborators: Hospital Universitario de la Plana (Other)
Responsible Party: Sponsor-Investigator, Marian Daras, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: MAR-ROP-2015-01
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Labor Epidural Analgesia
Keywords: epidural local anesthetic; epidural analgesia; analgesia labor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- IC+PIEB+PCEA high flow: Continuous Epidural Infusion to 3ml/h more Programed Intermittent Epidural Boluses of 7ml every hour with PCEA of 5 ml (interval of closing of 20min and maximum dose for hour of 15ml) administered with system of infusion of high flow as clinical practice routine
  Interventions: Device: IC+PIEB+PCEA high flow
- PIEB+PCEA high flow: Programed Intermittent Epidural Boluses of 10ml every hour with PCEA of 5 ml (interval of closing of 20min and maximum dose for hour of 15ml) administered with system of infusion of high flow as clinical practice routine
  Interventions: Device: PIEB+PCEA high flow
- PIEB+PCEA standar flow: Programed Intermittent Epidural Boluses of 10ml every hour with PCEA of 5 ml (interval of closing of 20min and maximum dose for hour of 15ml) administered with system of infusion of standar flow as clinical practice routine
  Interventions: Device: PIEB+PCEA standar flow

INTERVENTIONS:
Device: IC+PIEB+PCEA high flow — Ropivacaina 0,1 % is used with fentanilo 2ug/ml Also if during the dilation period a greater or equal AVE appears to 4 (inadequate analgesia) the patient can be administered a bolus of PCEA of the same solution.
  If the patient is administered PCEA, the programed intermittent epidural bolus is delayed automatically 20 minutes with regard to the time in which it would have to be administrated.
  If after two bolus of PCEA the analgesia keeps on being ineffective a clinical bolus is administered by the anaesthetist of 4ml of lidocaína to 1 %.
  This intervention is included in the clinical practice routine
  Groups: IC+PIEB+PCEA high flow
Device: PIEB+PCEA high flow — Ropivacaina 0,1 % is used with fentanilo 2ug/ml Also if during the dilation period a greater or equal AVE appears to 4 (inadequate analgesia) the patient can be administered a bolus of PCEA of the same solution.
  If the patient is administered PCEA, the programed intermittent epidural bolus is delayed automatically 20 minutes with regard to the time in which it would have to be administrated.
  If after two bolus of PCEA the analgesia keeps on being ineffective a clinical bolus is administered by the anaesthetist of 4ml of lidocaína to 1 %.
  In the group of pure boluses 10ml / h of perfusion will be administered through the high flow and standard flow infusion system, and the maximum sensory level achieved will be compared.
  This intervention is included in the clinical practice routine
  Groups: PIEB+PCEA high flow
Device: PIEB+PCEA standar flow — Ropivacaina 0,1 % is used with fentanilo 2ug/ml Also if during the dilation period a greater or equal AVE appears to 4 (inadequate analgesia) the patient can be administered a bolus of PCEA of the same solution.
  If the patient is administered PCEA, the programed intermittent epidural bolus is delayed automatically 20 minutes with regard to the time in which it would have to be administrated.
  If after two bolus of PCEA the analgesia keeps on being ineffective a clinical bolus is administered by the anaesthetist of 4ml of lidocaína to 1 %.
  In the group of pure boluses 10ml / h of perfusion will be administered through the high flow and standard flow infusion system, and the maximum sensory level achieved will be compared.
  This intervention is included in the clinical practice routine
  Groups: PIEB+PCEA standar flow

SUMMARY:
The investigators have design an observational study to know the anesthetic consumption in terms of rescue analgesia (Patient Controlled Epidural Analgesia (PCEA) and manual boluses) of the combination of different modes of administration of local anesthetic in the epidural space during labor analgesia offered by the new version of the CADD® infusion pump.

Also in this pump the anesthetic can be administered across a system of standard flow (40-250ml/h) or of high flow (40-500ml/h), what according to studies can influence the diffusion epidural of the anesthetic and therefore the level of sensitive blockade.

DETAILED DESCRIPTION:
The study is designed with healthy patients, first-time mothers, in childbearing dynamics, term pregnancy and nullipary. The epidural technique was performed with dose test of 3ml of bupivacaína 0,25 % with vasoconstrictor and a manual bolus of 0,1ml/Kg of ropivacaína 0,2% with fentanilo 5ug/ml.

As soon as the informed consent about the epidural anesthesia was signed, the patient was informed of the possibility of taking part in the study and there is offered him the sheet of information of the patient. So in one group they were administered Programed Intermittent Epidural Boluses (PIEB) and in other group continuous Epidural Infusion (IC) plus PIEB according to the usual clinical practice of each anesthesiologist. In both cases the perfusion was of ropivacaína 0,1 % more fentanilo 2ug/ml, so that in the first group it was administered PIEB of 10ml every hour and in the second group a continuous infusion to 3ml/h plus PIEB of 7ml every hour. Also if during the period of dilatation an AVE (Analogical Visual Escale) greater than or equal to 4 appeared (inadequate analgesia) the patient could administer a 5ml PCEA bolus of the same solution (interval of closing of 20min and maximum dose for hour of 15ml), as it is done in according to the usual clinical practice. And if after two boluses of PCEA the analgesia was still ineffective a clinical bolus of 4ml of lidocaína to 1 % was administered by the anesthesiologist.

In addition, in the group that was administered only PIEB, the standard infusion system was compared with the high-flow infusion system.

In all patients it was evaluated and noted on the epidural record sheet the intensity of the pain as the analogical visual scale (AVE), the grade of motor blockade as the modified scale of Bromage and the sensitive level in different periods of time. Also registered the total doses of anesthetic, the way of the childbearing finishes, the Apgar of the newborn, the grade of maternal satisfaction and the side effects. Also through the software of the pump it was verified if the patient had been administered rescue analgesia (PCEA or clinical boluses).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in work of established labor and contractions of moderate intensity
* Age between 18 and 45 years
* ASA I and II
* Nulliparity
* Pregnancy to term (> 36semanas)
* The only fetus of cephalic presentation
* Cervical dilation between 2-5cm

Exclusion Criteria:

* Maternal systemic illness (Diabetes Mellitus, arterial Hypertension, Preeclampsia. . )
* Major or equal weight to 100 Kg
* Less height of 150cm
* Duration of the equal or major childbearing to 24h
* Administration of opioides parenterales in 2-4h before to performing of the epidural
* Contraindication for neuroaxial analgesia
* Precedents of allergy or hypersensitivity to anesthetic local

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study will be realized in women in work of labor who come our hospital and who after being valued by the team of obstetrics are in favorable active period for the achievement of the technique epidural previous informed consent.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2015-08-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
anesthetic consumption in milliliters | at the end of labour
  The anesthetic consumption in terms of analgesia of rescue of the combination of different ways of administration of anesthetic in the space epidural. The quantity of extra analgesic is already by means of boluses of PCEA or by means of clinical boluses measured in milliliters

SECONDARY OUTCOMES:
analgesic effectiveness with AVE | Baseline (just after epidural administration)
  Measurement by means of the evaluation of the intensity of the pain that will be evaluated according to the analogical visual scale (AVE) with values between 0 and 10
analgesic effectiveness with AVE | 15 minutes after epidural administration
  Measurement by means of the evaluation of the intensity of the pain that will be evaluated according to the analogical visual scale (AVE) with values between 0 and 10
analgesic effectiveness with AVE | 30 minutes after epidural administration
  Measurement by means of the evaluation of the intensity of the pain that will be evaluated according to the analogical visual scale (AVE) with values between 0 and 10
analgesic effectiveness with AVE | every 2 hours until the end of labor
  Measurement by means of the evaluation of the intensity of the pain that will be evaluated according to the analogical visual scale (AVE) with values between 0 and 10
Motor blockade from zero to four | Baseline (just after epidural administration)
  The grade of motive blockade registers according to the modified scale of Bromage (from 0 to 3):
  0 = it can raise the low extremities of the bed
  1. = it can bend knees and ankles
  2. = it can bend ankles but not the knees
  3. = it can bend neither ankles nor knees
Motor blockade from zero to four | 15 minutes after epidural administration
  The grade of motive blockade registers according to the modified scale of Bromage (from 0 to 3):
  0 = it can raise the low extremities of the bed
  1. = it can bend knees and ankles
  2. = it can bend ankles but not the knees
  3. = it can bend neither ankles nor knees
Motor blockade from zero to four | 30 minutes after epidural administration
  The grade of motive blockade registers according to the modified scale of Bromage (from 0 to 3):
  0 = it can raise the low extremities of the bed
  1. = it can bend knees and ankles
  2. = it can bend ankles but not the knees
  3. = it can bend neither ankles nor knees
Motor blockade from zero to four | every 2 hours until the end of labor
  The grade of motive blockade registers according to the modified scale of Bromage (from 0 to 3):
  0 = it can raise the low extremities of the bed
  1. = it can bend knees and ankles
  2. = it can bend ankles but not the knees
  3. = it can bend neither ankles nor knees
Sensitive blockade from T12 to T4 | Baseline (just after epidural administration)
  The sensory level reached will be valued according to the loss of sensibility to the cold by means of a cotton with alcohol, noting down the dermatoma where it does not exist or diminishes the sensibility (T4: nipples level, T10: level of the bellybutton, T12: groin region). For statistical analysis of this variable a numerical value was given to each dermatome so that the highest value represents a higher sensory level and therefore more dermatomes with sensitive block (T12 = 0 and T4 = 8).
Sensitive blockade from T12 to T4 | 15 minutes after epidural administration
  The sensory level reached will be valued according to the loss of sensibility to the cold by means of a cotton with alcohol, noting down the dermatoma where it does not exist or diminishes the sensibility (T4: nipples level, T10: level of the bellybutton, T12: groin region ). For statistical analysis of this variable a numerical value was given to each dermatome so that the highest value represents a higher sensory level and therefore more dermatomes with sensitive block (T12 = 0 and T4 = 8).
Sensitive blockade from T12 to T4 | 30 minutes after epidural administration
  The sensory level reached will be valued according to the loss of sensibility to the cold by means of a cotton with alcohol, noting down the dermatoma where it does not exist or diminishes the sensibility (T4: nipples level, T10: level of the bellybutton, T12: groin region). For statistical analysis of this variable a numerical value was given to each dermatome so that the highest value represents a higher sensory level and therefore more dermatomes with sensitive block (T12 = 0 and T4 = 8).
Sensitive blockade from T12 to T4 | every 2 hours until the end of labor
  The sensory level reached will be valued according to the loss of sensibility to the cold by means of a cotton with alcohol, noting down the dermatoma where it does not exist or diminishes the sensibility (T4: nipples level, T10: level of the bellybutton, T12: groin region). For statistical analysis of this variable a numerical value was given to each dermatome so that the highest value represents a higher sensory level and therefore more dermatomes with sensitive block (T12 = 0 and T4 = 8).
Blood pressure | Baseline (just after epidural administration)
  The patient will be evaluated and there will register the blood pressure in mm of mercury
Blood pressure | 15 minutes after epidural administration
  The patient will be evaluated and there will register the blood pressure in mm of mercury
Blood pressure | 30 minutes after epidural administration
  The patient will be evaluated and there will register the blood pressure in mm of mercury
Blood pressure | every 2 hours until the end of labor
  The patient will be evaluated and there will register the blood pressure in mm of mercury
Maternal heart rate | Baseline (just after epidural administration)
  The patient will be evaluated and there will register the maternal heart rate in beats per minute
Maternal heart rate | 15 minutes after epidural administration
  The patient will be evaluated and there will register the maternal heart rate in beats per minute
Maternal heart rate | 30 minutes after epidural administration
  The patient will be evaluated and there will register the maternal heart rate in beats per minute
Maternal heart rate | every 2 hours until the end of labor
  The patient will be evaluated and there will register the maternal heart rate in beats per minute
maternal satisfaction | at the end of labor
  On having finished the childbearing, from 0 to 100 will value the grade of maternal satisfaction as an evaluation scale:
  * 0 = very unsatisfied with the analgesia provided by the treatment
  * 100 = extremely satisfied with the analgesia provided by the treatment
adverse effects | at the end of labor
  There will be noted down also the appearance of adverse effects as the sickness and vomiting, urinal retention, pruritus and fever.

OTHER OUTCOMES:
Weight in kilograms | Just before epidural administration
  The weight in kilograms will be noted on the epidural record sheet
Size in centimeters | Just before epidural administration
  The height in centimeters will be noted on the epidural record sheet
ASA from one to five | Just before epidural administration
  The ASA classification will be noted on the epidural record sheet
Gestational week in number | Just before epidural administration
  The Gestational week in number will be noted on the epidural record sheet
Cervical dilatation at the time of performing the epidural technique in centimeters | Just before epidural administration
  The dilatation in centimeters will be noted on the epidural record sheet
Administration of parenteral opioids and the time of administration | Just before epidural administration
  In the epidural record sheet if opioids have been administered it will be recorded as YES and if they have not been administered it will be recorded as NO. If it has been administered, the time of its admnistracion will be indicated numerically

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Plana, Villarreal, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albright GA, Forster RM. The safety and efficacy of combined spinal and epidural analgesia/anesthesia (6,002 blocks) in a community hospital. Reg Anesth Pain Med. 1999 Mar-Apr;24(2):117-25. doi: 10.1016/s1098-7339(99)90071-8. PMID 10204896
- [Background] Beaubien G, Drolet P, Girard M, Grenier Y. Patient-controlled epidural analgesia with fentanyl-bupivacaine: influence of prior dural puncture. Reg Anesth Pain Med. 2000 May-Jun;25(3):254-8. doi: 10.1016/s1098-7339(00)90007-5. PMID 10834779
- [Background] Simmons SW, Taghizadeh N, Dennis AT, Hughes D, Cyna AM. Combined spinal-epidural versus epidural analgesia in labour. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003401. doi: 10.1002/14651858.CD003401.pub3. PMID 23076897
- [Background] Patel NP, El-Wahab N, Fernando R, Wilson S, Robson SC, Columb MO, Lyons GR. Fetal effects of combined spinal-epidural vs epidural labour analgesia: a prospective, randomised double-blind study. Anaesthesia. 2014 May;69(5):458-67. doi: 10.1111/anae.12602. PMID 24738803
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Background] Birnbach DJ, Ojea LS. Combined spinal-epidural (CSE) for labor and delivery. Int Anesthesiol Clin. 2002 Fall;40(4):27-48. doi: 10.1097/00004311-200210000-00005. No abstract available. PMID 12409932
- [Background] Polley LS, Columb MO, Naughton NN, Wagner DS, van de Ven CJ. Relative analgesic potencies of ropivacaine and bupivacaine for epidural analgesia in labor: implications for therapeutic indexes. Anesthesiology. 1999 Apr;90(4):944-50. doi: 10.1097/00000542-199904000-00003. PMID 10201661
- [Background] Johnson RF, Cahana A, Olenick M, Herman N, Paschall RL, Minzter B, Ramasubramanian R, Gonzalez H, Downing JW. A comparison of the placental transfer of ropivacaine versus bupivacaine. Anesth Analg. 1999 Sep;89(3):703-8. doi: 10.1097/00000539-199909000-00032. PMID 10475309
- [Background] Beilin Y, Guinn NR, Bernstein HH, Zahn J, Hossain S, Bodian CA. Local anesthetics and mode of delivery: bupivacaine versus ropivacaine versus levobupivacaine. Anesth Analg. 2007 Sep;105(3):756-63. doi: 10.1213/01.ane.0000278131.73472.f4. PMID 17717236
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Carvalho B, George RB, Cobb B, McKenzie C, Riley ET. Implementation of Programmed Intermittent Epidural Bolus for the Maintenance of Labor Analgesia. Anesth Analg. 2016 Oct;123(4):965-71. doi: 10.1213/ANE.0000000000001407. PMID 27464978
- [Background] Epsztein Kanczuk M, Barrett NM, Arzola C, Downey K, Ye XY, Carvalho JC. Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Biased-Coin Up-and-Down Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 10 mL of Bupivacaine 0.0625% With Fentanyl 2 mug/mL. Anesth Analg. 2017 Feb;124(2):537-541. doi: 10.1213/ANE.0000000000001655. PMID 27755057
- [Background] Delgado C, Ciliberto C, Bollag L, Sedensky M, Landau R. Continuous epidural infusion versus programmed intermittent epidural bolus for labor analgesia: optimal configuration of parameters to reduce physician-administered top-ups. Curr Med Res Opin. 2018 Apr;34(4):649-656. doi: 10.1080/03007995.2017.1377166. Epub 2017 Oct 6. PMID 28875709
- [Background] Sng BL, Zeng Y, de Souza NNA, Leong WL, Oh TT, Siddiqui FJ, Assam PN, Han NR, Chan ES, Sia AT. Automated mandatory bolus versus basal infusion for maintenance of epidural analgesia in labour. Cochrane Database Syst Rev. 2018 May 17;5(5):CD011344. doi: 10.1002/14651858.CD011344.pub2. PMID 29770432
- [Background] Klumpner TT, Lange EM, Ahmed HS, Fitzgerald PC, Wong CA, Toledo P. An in vitro evaluation of the pressure generated during programmed intermittent epidural bolus injection at varying infusion delivery speeds. J Clin Anesth. 2016 Nov;34:632-7. doi: 10.1016/j.jclinane.2016.06.017. Epub 2016 Aug 3. PMID 27687462
- [Background] Krawczyk P, Piwowar P, Salapa K, Lonc T, Andres J. Do Epidural Catheter Size and Flow Rate Affect Bolus Injection Pressure in Different Programmed Intermittent Epidural Bolus Regimens? An In Vitro Study. Anesth Analg. 2019 Dec;129(6):1587-1594. doi: 10.1213/ANE.0000000000003650. PMID 31743179
- [Result] Loubert C, Hinova A, Fernando R. Update on modern neuraxial analgesia in labour: a review of the literature of the last 5 years. Anaesthesia. 2011 Mar;66(3):191-212. doi: 10.1111/j.1365-2044.2010.06616.x. PMID 21320088